CLINICAL TRIAL: NCT02823821
Title: Randomised Evaluation of Sodium Dialysate Levels on Vascular Events
Acronym: RESOLVE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australasian Kidney Trials Network (Network); Australia & New Zealand Dialysis & Transplant Registry (Unknown); The George Institute (Other); The George Institute for Global Health, China (Other); Peking University People's Hospital (Other); Institute for Clinical Evaluative Sciences (Other); St. Michaels Hospital (Unknown); University Hospital Wuerzburg, Medizinische Klinik EINS (Unknown); Malaysian Society of Nephrology (Unknown); Malaysian Renal Registry (Unknown); Comprehensive Clinical Trials Unit, University College London (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GI-AU-RM-2016-01
Record Dates: First submitted 2016-06-16; First posted 2016-07-06 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: End-Stage Kidney Disease
Keywords: End-Stage Kidney Disease; Hemodialysis; Dialysate; Sodium; Cluster-randomisation; Dialysis; RESOLVE
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 137mmol/l (Active Comparator): Participating dialysis sites will be randomised to a default dialysate sodium concentration of 137mmol/l
  Interventions: Other: Default dialysate sodium concentration of 137mmol/l
- 140mmol/l (Active Comparator): Participating dialysis sites will be randomised to a default dialysate sodium concentration of 140mmol/l
  Interventions: Other: Default dialysate sodium concentration of 140mmol/l

INTERVENTIONS:
Other: Default dialysate sodium concentration of 137mmol/l — Default defined here as use of allocated dialysate sodium concentration for at least 90% of delivered dialysis sessions.
  Arms: 137mmol/l
Other: Default dialysate sodium concentration of 140mmol/l — Default defined here as use of allocated dialysate sodium concentration for at least 90% of delivered dialysis sessions.
  Arms: 140mmol/l

SUMMARY:
This global study will assess the effect of randomising dialysis sites to one of two default dialysate sodium concentrations in current practice, 140mmol/l and 137mmol/l, on major cardiovascular events and death in patients receiving maintenance haemodialysis.

DETAILED DESCRIPTION:
RESOLVE is a pragmatic, cluster-randomised, open-label study designed to evaluate in real-world conditions the comparative effectiveness of two default dialysate sodium concentrations.

Dialysis sites will be randomised in a 1:1 ratio to a default dialysate sodium concentration of 137mmol/l or 140mmol/l. 'Default' is defined as the use of the allocated dialysate sodium for ≥ 90% of delivered dialysis sessions in the unit. All other care will be according to standard local practices as determined by the site.

Outcomes will be assessed on individual patients dialysing at those sites. Sites will be asked to consent to participation while waiver or opt-out consent will be sought for individual patients.

It is anticipated that site accrual will occur over 5-7 years with average study duration expected to be approximately 2-5 years. The actual length of the study will be end-point determined.

ELIGIBILITY:
The site inclusion criteria are:

* Predominantly dialyses adults (≥18 years old) receiving maintenance haemodialysis
* Rates of withdrawal within the first two years of commencing dialysis for social reasons have been less than 15% for the 2 years prior to recruitment and are not expected to increase above 15%
* Has a minimum of 10 dialysis recipients at time of randomisation
* Utilises a default dialysate sodium concentration at the time of recruitment (a substantial majority of dialysis sessions are conducted with the default dialysate sodium concentration)
* Is a self-contained unit (i.e. unit patients do not regularly rotate through another unit. Brief trips by patients to a parent or other unit do not exclude a site)
* Willing to accept randomisation to either intervention (as determined by nominated Director of Unit)
* Is not a home dialysis training or support unit. [Sites that include both in-center/satellite dialysis patients and home patients may participate but the study procedures and assessments will only be conducted in the incenter/satellite component of the site].

The exclusion criteria are:

* Not able to comply with data collection methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of an event in the primary composite outcome | Through to study completion (estimated to occur after an average of 5 years follow up)
  Primary outcome is a composite of major cardiovascular events (hospitalised acute myocardial infarction, hospitalised stroke) and all-cause death. Study completion is endpoint driven, but is expected to be when the average follow up is around 5 years.

SECONDARY OUTCOMES:
Time to first occurrence of an event in the secondary composite outcome | Through to study completion (estimated to occur after an average of 5 years follow up)
  Secondary outcome comprises major cardiovascular events (hospitalized acute myocardial infarction, hospitalized stroke), all-cause death and hospitalized heart failure. Study completion is endpoint driven, but is expected to be when the average follow up is around 5 years.
Time to first occurrence of each of the individual components of the composite outcomes. | Through to study completion (estimated to occur after an average of 5 years follow up)
  These components are hospitalised myocardial infarctions, hospitalised strokes, hospitalised heart failures and all-cause deaths. Study completion is endpoint driven, but is expected to be when the average follow up is around 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Meg Jardine, Study Director — The University of Sydney, NHMRC Clinical Trials Centre; Carmel Hawley, Study Chair — The University of Queensland; Vivekanand Jha, Study Chair — The George Institute India; Zuo Li, Study Chair — Peking University People's Hospital; Sunita Bavanandan, Study Chair — Kuala Lumpur General Hospital; David Wheeler, Study Chair — Comprehensive Clinical Trials Unit, University College London; Patrick Rossignol, Study Chair — INSERM Clinical Investigation Centre; Mike Walsh, Study Chair — McMaster University; Vlado Perkovic, Study Chair — University of New South Wales; Christoph Wanner, Study Chair — University Hospital Wuerzburg; Jule Pinter, Principal Investigator — University Hospital Wuerzburg
Locations (264):
- Australia (31):
  - Royal Adelaide Hospital, Adelaide
  - Auburn Hospital, Auburn
  - Flinders Medical Centre, Bedford Park
  - Moorabbin Hospital, Bentleigh East
  - Sunshine Coast University Private Hospital, Birtinya
  - Princess Alexandra Hospital, Brisbane
  - Redlands Hospital, Brisbane
  - Bundaberg Hospital, Bundaberg
  - Caloundra Hospital, Caloundra
  - Royal Prince Alfred Hospital, Camperdown
  - The Canberra Hospital, Canberra
  - Peninsula Health, Frankston
  - Gympie Hospital, Gympie
  - Ipswich Hospital, Ipswich
  - Mackay Base Hospital, Mackay
  - Logan Hospital, Meadowbrook
  - Monash Health Community Dandenong, Melbourne
  - Casey Hospital, Melbourne
  - Cranbourne Integrated Care Centre, Melbourne
  - Nambour General Hospital, Nambour
  - Hampstead Dialysis Centre, Northfield
  - Hervey Bay Hospital, Pialba
  - Royal North Shore Hospital, St Leonards
  - Sunshine Coast University Hospital, Sunshine Coast
  - Sydney Adventist Hospital, Sydney
  - Concord Repatriation and General Hospital, Sydney
  - Blacktown Regional Dialysis Centre, Sydney
  - Mt Druitt Community Dialysis Centre, Sydney
  - Nepean Hospital, Sydney
  - Westmead Hospital, Sydney
  - The Queen Elizabeth Hospital, Woodville South
- Canada (20):
  - Brantford General Hospital, Brantford, Ontario
  - Chatam-Kent Health Alliance, Chatham, Ontario
  - St Joseph's Healthcare, Hamilton, Ontario
  - Hanover District Hospital, Hanover, Ontario
  - Adam Linton Dialysis Unit - Victoria Hospital, London, Ontario
  - London Health Sciences Centre, London, Ontario
  - Westmount Kidney Care Centre, London, Ontario
  - Grey Bruce Health Services, Owen Sound, Ontario
  - Bluewater Hospital, Sarnia, Ontario
  - Huron Perth Hospital Partnership, Stratford, Ontario
  - Tillsonburg District Memorial Hospital, Tillsonburg, Ontario
  - Woodstock General Hospital, Woodstock, Ontario
  - Stoney Creek, Hamilton
  - Belleville, Kingston
  - Brockville, Kingston
  - Kingston General, Kingston
  - Napanee, Kingston
  - Perth and Smith Falls, Kingston
  - Picton, Kingston
  - St. Michael's Hospital, Toronto
- Germany (16):
  - Nephrologisches Zentrum Albstadt, Albstadt
  - Praxis für Nierenkrankheiten Berlin Hellersdorf, Berlin
  - Dialyse am Kortumpark Bochum, Bochum
  - Dialysezentrum Darmstadt, Darmstadt
  - Dialysezentrum Elsenfeld, Elsenfeld
  - Nephrologisches Zentrum Hechingen, Hechingen
  - Arbeitsgemeinschaft Heimdialyse Saar e.V., Homburg
  - Dialysezentrum Langen, Langen
  - KfH Nierenzentrum Lichtenfels, Lichtenfels
  - Universitätsmedizin Mainz, Dialysestation 605-5E, Mainz
  - KfH Nierenzentrum München Schwabing, Munich
  - UBAG Öhringen, Öhringen
  - Dialysezentrum Schweinfurt, Schweinfurt
  - Dialysezentrum Siegburg, Siegburg
  - Nephrologie - Dialyse - Christliches Klinikum Unna, Unna
  - Nephrologisches Zentrum Villingen-Schwenningen -Tuttlingen, Villingen-Schwenningen
- India (63):
  - Area Hospital, Kothapeta Road,Chirala, Andhra Pradesh, Chīrāla, Andhra Pradesh
  - Government General Hospital, Guntur, Andhra Pradesh
  - Medical Superintendent Government Hospital, Gūdūr, Andhra Pradesh
  - Medical Superintendent District Hospital, Hindupur PPP, Andhra Pradesh
  - Government Area Hospital, Kanigiri, Andhra Pradesh, Kanigiri, Andhra Pradesh
  - Government Hospital, Kākināda, Andhra Pradesh
  - Government General Hospital, Kurnool, Andhra Pradesh
  - Government Hospital, Machilipatnam PPP, Andhra Pradesh, Machilipatnam, Andhra Pradesh
  - Government Area Hospital, Mārkāpur, Andhra Pradesh
  - Government Hospital, Nandyāl, Andhra Pradesh
  - Area Hospital, Narsīpatnam, Andhra Pradesh
  - Government Area Hospital, Palakonda, Srikakulam District, Andhra Pradesh
  - CHC Government Hospital, Palāsa, Andhra Pradesh
  - Government Area Hospital, Pārvathipuram, Andhra Pradesh
  - Government Hospital, Proddatūr, Andhra Pradesh
  - Government Hospital, Rajahmundry, Andhra Pradesh
  - CHC Hospital, Sompeta, Andhra Pradesh, Sompeta, Andhra Pradesh
  - Greater Kailash Hospital, Tadepalligudem, Andhra Pradesh
  - Manasa Kidney Foundation, Tirupati, Andhra Pradesh
  - Government General Hospital, Vijayavada PPP, Andhra Pradesh, Vijayawada, Andhra Pradesh
  - King George Government Hospital, Visakhapatnam, Andhra Pradesh
  - Ford Hospital, Khemnichak, Patna, Patna, Bihar
  - Janak Dulari Hospital, Hanuman Nagar, Patna, Bihar
  - Aysha Hospital, Kilpauk, Chennai
  - Retteri Sri Kumaran Health Centre, Kolathūr, Chennai
  - Leelawati Hospital, Ambāla, Haryana
  - Greater Kailash Hospital, Old Palasia, Indore
  - ESI Hospital, Bhetia, Jharkand
  - K.M Memorial Hospital and Research Centre, Bokāro, Jharkhand
  - Asarfi Hospital, Dhanbad, Jharkhand
  - Bhagwan Mahavir Medical Superspeciality Hospital, Ranchi, Jharkhand
  - Guru Nanak Hospital and Research Centre, Ranchi, Jharkhand
  - Koshys Hospital, Ramamurthy Nagar, Bengaluru, Karnataka
  - Nephroplus Basaveshwaranagar, Bengaluru, Karnataka
  - Fortis Suchirayu Hospital, Hubli, Karnataka
  - Main Hospital, SCCL, Kothagudem, Khammam
  - Vishesh Hospital Pvt. Ltd, Geeta Bhawan Chouraha, Indore, Madhya Pradesh
  - Hitwardhak Mandal Hospital, Mumbai, Maharashtra
  - Lokmanya Hospital, Pune, Maharashtra
  - Chirayu Hospital, Thane, Maharashtra
  - Nephroplus Borivali Standalone, Borivali West, Mumbai
  - Bharat Baug, Borivali West, Mumbai
  - Jyothi Hospital, Balasore, Odisha
  - Kar Clinic & Hospital Pvt. Ltd., Bhubaneswar, Odisha
  - Neelachal Hospital, Kharvel Nagar, Bhubaneswar, Odisha
  - Satguru Partap Singh Apollo Hospitals, Ludhiana, Punjab
  - Deepam Hospitals, Pallavaram, Chennai, Tamil Nadu
  - KG Hospital, Coimbatore, Tamil Nadu
  - Neyveli Lignite Corporation Hospital, Neyveli, Tamil Nadu
  - Sudha Hospital, Vadalur, Neyveli, Tamil Nadu
  - Citizens Specialty Hospital, Hyderabad, Telangana
  - ESI Multi-Specialty Hospital, Hyderabad, Telangana
  - Vintage Plaza Nephroplus, Road no. 10, Banjara Hills, Hyderabad, Telangana
  - Government Hospital, Khammam, Telangana
  - Suraksha Multispecialty Hospital, Nalgonda, Telangana
  - Nephroplus Standalone Dialysis Center, Easy Marredpally, Secunderabad, Telangana
  - Rajiv Gandhi Institute of Medical Sciences, Srikakulam PPP, Andhra, Srikakulam, Telangana
  - Madhuraj Hospital, Kanpur, Uttar Pradesh
  - Ajanta Hospital, Lucknow, Uttar Pradesh
  - Surbhi Hospital Pvt. Ltd, Sector 35, Noida, Uttar Pradish
  - Health Point Hospital, Prannth Pandit Street, Kolkata, West Bengal
  - Minimal Access Surgery Clinic Pvt Ltd, Tamlūk, West Bengal
  - Baroma Sirona Hospital, Uttar Mechgram, West Bengal
- Malaysia (39):
  - Hospital Ampang, Ampang
  - Hospital Sultanah Nora Ismail, Batu Pahat
  - Hospital Beaufort, Beaufort
  - Hospital Pulau Pinang, George Town
  - Pusat Dialisis NKF- Yayasan Dialisis Pendidikan Akhlak Perak, Ipoh
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Kajang, Kajang
  - Hospital Serdang, Kajang
  - Hospital Tuanku Fauziah, Kangar
  - Pusat Rawatan Dialisis Tuanku Syed Putra - NKF, Kangar
  - Hospital Tengku Ampuan Rahimah, Klang
  - Pusat Daillisis NKF - Kelab Apex, Klang
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Hospital Likas, Kota Kinabalu
  - Hospital Queen Elizabeth II, Kota Kinabalu
  - Hospital Kuala Kangsar, Kuala Kangsar
  - Hospital Kuala Lipis, Kuala Lipis
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pusat Dialisis NKF-Fungates Superflow, Kuala Lumpur
  - Pusat Dialisis NKF-Nanyang, Kuala Lumpur
  - Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Kudat, Kudat
  - Hospital Kulim, Kulim
  - Hospital Labuan, Labuan
  - Hospital Sultanah Bahiyah, Langgar
  - Haemodialysis Unit Klinik Kesihatan Lenggong, Lenggong
  - Pusat Hemodialisis Komuniti Cheng, Malacca
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Hospital Seberang Jaya, Permatang Pauh
  - Pusat Dialisis NKF - Chempaka, Petaling Jaya
  - Hospital Shah Alam, Shah Alam
  - Universiti Teknologi Mara, Shah Alam
  - Hospital Sultan Abdul Halim, Sungai Petani
  - Hospital Sungai Siput, Sungai Siput
  - Hospital Tambunan, Tambunan
  - Hospital Sultan Haji Ahmad Shah, Temerluh
- United Kingdom (95):
  - Altrincham General Hospital Dialysis Unit, Altrincham
  - Tameside Renal Dialysis Unit, Ashton-under-Lyne
  - Barnet Satellite Unit, Barnet
  - Barnsley Dialysis Unit, Barnsley
  - Bath Dialysis Unit, Bath
  - Bedford Renal Unit, Bedford
  - Bexhill Dialysis Unit, Bexhill-on-Sea
  - Hexagon Towers Dialysis Unit, Blackley
  - Bolton Kidney Care Centre, Bolton
  - St Luke's Hospital Renal Ward, Bradford
  - Bridgwater Dialysis Unit, Bridgwater
  - Brighton Sussex Kidney Unit, Brighton
  - Cossham Dialysis Unit, Bristol
  - South Bristol Dialysis Unit, Bristol
  - Bromley Dialysis Unit, Bromley
  - Broomfield Hospital, Broomfield
  - Cannock Haemodialysis Unit, Cannock
  - Chesterfield Dialysis Unit, Chesterfield
  - Clacton (Diaverum), Clacton-on-Sea
  - Colchester (Diaverum), Colchester
  - Clay Lane, Coventry
  - University Hospitals Coventry & Warwickshire Main Unit, Coventry
  - Crawley Dialysis Unit, Crawley
  - Leighton, Crewe
  - Cromer Hospital Dialysis Unit, Cromer
  - Darlington Dialysis Unit, Darlington
  - Dartford Dialysis Unit, Dartford
  - Dover Renal Unit, Dover
  - Edgware Satellite Unit, Edgware
  - Epsom Dialysis Unit, Epsom
  - Heavitree, Exeter
  - Farnborough Dialysis Unit, Farnborough
  - Cotswold Dialysis Centre, Gloucester
  - Severn, Gloucester
  - James Paget Renal Unit, Great Yarmouth
  - Grimsby Renal Unit, Grimsby
  - Harlow Renal Unit, Harlow
  - Hayes Hospital, Hayes
  - Honiton, Honiton
  - Chiltern Renal Unit, Houghton Regis
  - Fresenius Hull Dialysis Unit, Hull
  - West Middlesex, Isleworth
  - Kingston Satellite Dialysis Unit, Kingston
  - Collierswood Dialysis Unit, London
  - King George Hospital, London
  - Mary Rankin Satellite Unit, London
  - North Wandsworth Dialysis Unit, London
  - Royal London Hospital, London
  - Whipps Cross Hospital, London
  - Ludlow Dialysis Unit, Ludlow
  - Macclesfield District General Hospital, Macclesfield
  - Manchester Royal Infirmary Renal Dialysis Unit, Manchester
  - Octagon Renal Satellite, Manchester
  - Margate Renal Unit, Margate
  - James Cook, Middlesbrough
  - North Ormesby, Middlesbrough
  - Harrogate, North Yorks
  - Friarage Hospital, Northallerton
  - Lucy Deane (George Eliot), Nuneaton
  - Oldham Dialysis Unit, Oldham
  - Newham Hospital, Plaistow
  - Eastbourne (Polegate) Dialysis Unit, Polegate
  - Rochdale Dialysis Unit, Rochdale
  - Queen's Hospital, Romford
  - Rotherham Dialysis Unit, Rotherham
  - St Cross (Ash Unit), Rugby
  - Salford Renal Unit, Salford
  - Scarborough, Scarborough
  - Scunthorpe Dialysis Centre, Scunthorpe
  - Peter Moorhead Unit, Sheffield
  - Renal G Floor, Sheffield
  - Sheffield Dialysis Unit, Sheffield
  - Shrewsbury Renal Unit, Shrewsbury
  - Smethwick Dialysis Centre, Smethwick
  - St Albans Dialysis Unit, St Albans
  - County Hospital, Stafford
  - Lister Renal Unit, Stevenage
  - Stockport NHS Dialysis Unit, Stockport
  - North Tees, Stockton-on-Tees
  - Royal Stoke, Stoke-on-Trent
  - Stratford Dialysis Centre, Stratford-upon-Avon
  - St. Helier Dialysis Unit, Sutton
  - Sutton Dialysis Unit, Sutton
  - Taunton Dialysis Centre, Taunton
  - Hollinswood House Renal Unit, Telford
  - Croydon Dialysis Unit, Thornton Heath
  - South Devon Satellite Kidney Unit, Torquay
  - Tottenham Hale Satellite Unit, Tottenham
  - Wigan Renal Unit, Wigan
  - Ashford Renal Unit, Willesborough
  - Pond Lane Dialysis Unit, Wolverhampton
  - Woolwich Dialysis Unit, Woolwich
  - Worthing Dialysis Unit, Worthing
  - Easingwold, York
  - York Hospital, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinter J, Canaud B, Mayne KJ, Stuard S, Moissl U, Kooman J, Jager KJ, Chesnaye NC, Smyth B, Genser B. Associations of Abnormal Fluid Status, Plasma Sodium Disorders, and Low Dialysate Sodium with Mortality in Patients on Hemodialysis. Clin J Am Soc Nephrol. 2024 Nov 1;19(11):1444-1452. doi: 10.2215/CJN.0000000000000552. Epub 2024 Sep 10. PMID 39514693
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822
- [Derived] See EJ, Polkinghorne KR. Volume management in haemodialysis patients. Curr Opin Nephrol Hypertens. 2020 Nov;29(6):663-670. doi: 10.1097/MNH.0000000000000642. PMID 32889978